CLINICAL TRIAL: NCT07209592
Title: Effect of Artificial Intelligence Based Gamification Training on Cognition and Functional Outcomes in Patients With Stroke
Acronym: AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Rabee Shehab, principle investigator : mai rabee ahmed shehab, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005963
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Artificial Intelligence Based Gamification Training; Cognition; Functional Outcomes
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Artificial Intelligence Based Gamification Training and Exercise Program
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI gamification (Experimental): twenty patients will receive cognitive tasks accompanied by cognitive-driven motor tasks by AI gamification plus conventional therapy three times per weeks for four weeks
  Interventions: Other: AI gamification; Other: conventional therapy
- conventional therapy (Active Comparator): twenty patients will receive conventional therapy exercises three times per weeks for four weeks
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: AI gamification — The treatment program for AI gamification group will be in the form of cognitive tasks accompanied by cognitive driven motor tasks ( integrating cognitive strategies into motor tasks) exercises of the upper limb (shoulder, elbow, hand) in the form of AI gamification model. For each patient in study group, session will be for 6 minutes , three times per week for 4 weeks. The patients Will receive AI gamification via X-box with 3 D kinetic motion analysis giving the patient real time feedback, visual and auditory feedback about the range and task .Using this technology we will gain the benefits of both AI and Gamification, the patients will be engaged in the exercise intensively and for a longer time with out getting bored and the tasks will be enjoyable to capture their attention , in addition to traditional training plus conventional therapy
  Arms: AI gamification
Other: conventional therapy — the patiens will receive conventional therapy exercises in the form of flexibility exercises, strengthening exercises, Aerobic training exercise
  * flexibility exercises , it will be in the form of functional stretching for shoulder adductors and flexors, elbow flexors ,wrist and finger flexors
  * strengthening exercises , it will be mainly strengthening exercises for upper limb (shoulder extensors, elbow , wrist and finger extensors) in addition to trunk control exercises targeting proximal stability for distal mobility.
  Aerobic training exercise, as a form of cognitive training exercises

SUMMARY:
this study will be conducted to investigate the effect of artificial intelligence based gamification training on cognition and functional outcomes in patients with stroke

DETAILED DESCRIPTION:
Stroke is a neurological disorder characterized by blockage of blood vessels. Clots form in the brain and interrupt blood flow, clogging arteries and causing blood vessels to break, leading to bleeding. Rupture of the arteries leading to the brain during stroke results in the sudden death of brain cells owing to a lack of oxygen. Stroke can also lead to depression and dementia.Cognitive impairment refers to a broad range of deficits in cognitive function, including memory, attention, executive function, language, and visuo-spatial skills. Understanding the connection between stroke and cognitive impairment is crucial for effectively managing symptoms and improving stroke survivors' quality of life.Gamified interventions outperformed conventional therapies in reducing task, completion time , Sustained Engagement. AI-driven adaptive systems, such as the Bright Brainer Grasp (BBG) controller, increased patient motivation by dynamically adjusting difficulty levels based on real-time performance reducing caregiver oversight. BCI and Gamification Synergy , Brain-Computer Interface (BCI) systems combined with gamified tasks (e.g., CoWMeG) improved upper limb motor function. Motor Imagery: Enhanced neural plasticity through imagined movements .Mirror Neuron Activation: Visual feedback from avatars reinforced motor learning..Therefore this study will be designed to investigate the effect of gamification AI based training on cognition in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Forty hemiplegic patients with mild post stroke cognitive impairment.
* The patients age will be 45 to 60.
* Chronic stroke (6 months post-stroke).
* Score of 1 to 1+ to points on the Modified Ashworth Scale (MAS) on upper limb (shoulder , elbow ,hand).
* Stage of recovery 4-5 brunnstrom
* Essential educational level ( at least high school level)
* BMI will be ranged from 18,5 -24.9 kg\m2

Exclusion Criteria:

* Moderate and severe post stroke cognitive impairment
* Excluding cognitive impairment for any other psychological or neurological disease such as depression and dementia
* history of recent upper limb surgery
* Any musculoskeletal disorders of upper extremity (e.g fractures or injuries)
* Having a heart pacemaker, pregnancy
* Other neurological diseases or cancer
* Hormonal disturbances

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
cognitive disability | up to four weeks
  cognition will be measured by Smart phone- based cognitive assessement allows older adults to be more engaged in cognitive screening and monitoring both inside and outside the clinic. It provide advantages over the traditional cognitive testing such as cost ,time saving, more detailed response metric recordings, automated data collection and scoring.
upper limb function | up to four weeks
  Wolf Motor Functional scale will be used for assessment of upper limb function.The original version of the WMFT consisted of 21 items. The widely used version of the WMFT consists of 17 items .It is composed of three parts namely, time, functional ability (items 1-6) and strength (items 7-14). Remaining 9 items involves analysing movement quality when completing various tasks. The less affected side is tested first, followed by the affected limb. The following tasks should be completed as quickly as possible, with a 120-second time limit.
handgrip strength | up to four weeks
  A handheld dynamometer will be used for assessing hand grip strength
kinetic motion analysis | up to four weeks
  X - Box kinetic motion sensor devcie will be used for assessing motion analysis